CLINICAL TRIAL: NCT06911554
Title: A Phase III Clinical Study of Recombinant Human Albumin Injection for the Treatment of Hypoalbuminemia in Cirrhotic Patients With Ascites
Brief Title: A Study of Recombinant Human Albumin Injection to Treat Hypoalbuminemia in Cirrhotic Patients With Ascites
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tonghua Anrate Biopharmaceutical Co., Ltd. (Industry)
Collaborators: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ART-2021-005
Record Dates: First submitted 2025-03-25; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Hepatic Ascites
Keywords: Hepatic Ascites
MeSH Terms: interventions — Serum Albumin, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Experimental): Recombinant Human Albumin Injection, 20g/day, once daily for 7 days
  Interventions: Biological: Recombinant Human Albumin Injection
- Control group (Active Comparator): Human Albumin, 20g/day, once daily for 7 days
  Interventions: Biological: Human Albumin

INTERVENTIONS:
Biological: Recombinant Human Albumin Injection — Recombinant Human Albumin injection, strength: 10 g/vial (20%, 50 mL); storage conditions: 2-8°C, protected from light; manufactured and supplied by Tonghua Anrate Biopharmaceutical Co., Ltd.
  Arms: Treatment group
Biological: Human Albumin — Human Albumin (An Pu Lai Shi®), strength: 10 g/vial (protein concentration 20%, 50 mL/vial), storage conditions: 2-8°C, protected from light; manufactured by Shanghai RAAS Blood Products Co., Ltd.
  Arms: Control group

SUMMARY:
This study was a Phase III multicenter, blinded, and positive active-controlled clinical study to evaluate the efficacy, safety, and immunogenicity of recombinant human albumin(rHA) injection for the treatment of hypoalbuminemia in cirrhotic patients with ascites.

DETAILED DESCRIPTION:
This study was a Phase III multicenter, blinded, and positive active-controlled clinical study to evaluate the efficacy, safety, and immunogenicity of recombinant human albumin(rHA) injection for the treatment of hypoalbuminemia in cirrhotic patients with ascites.After the primary efficacy endpoint ALB reaches the equivalence standard (-2 g/L to 2 g/L, test drug - control drug), a non-inferiority judgment will be made for the key secondary efficacy endpoint of the improvement rate of ascites depth (> -10%, test drug - control drug). Dosage: 20 g/day once daily for 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18-75 years (inclusive）.
* BMI≥18.0 kg/m^2.
* Subjects who were diagnosed as liver cirrhosis with ascites according to the Guidelines for Diagnosis and Treatment of Liver Cirrhosis with Ascites and Related Complications (2017) issued by the Chinese Society of Hepatology CMA, with ascites graded 1-2 at diagnosis or after treatment, and also met the requirement of ALB < 30 g/L ;
* Subjects who were able to understand and comply with the study procedures, voluntarily participated this study, and had signed the informed consent form (ICF).

Exclusion Criteria:

* Subjects with a history of allergies to biological products derived from Escherichia coli, yeast, or Chinese hamster ovary (CHO) cells, or blood products such as HSA.
* Subjects with hepatic encephalopathy of West-Haven HE Grade III or higher.
* Subjects with uncontrolled infections, such as body temperature > 37.5°C, white blood cell count > 1.0 × 10^10/L, or severe abdominal infection, upper respiratory tract infection, lower respiratory tract infection, urinary system infection, etc.).
* Subjects with a history of hepatorenal syndrome (HRS), or serum creatinine (Cr) > 2 × the upper limit of normal (ULN), or Cr increased by > 50% during screening period; or presence of urine protein 2+ or more.
* Subjects with other severe underlying conditions that, in the opinion of the investigator, affected the participation in this study, including but not limited to malignancies (exclusion criteria below for liver cancer patients), complicated portal vein thrombosis, non-cirrhotic portal hypertension-related ascites, ischemic heart disease, stroke, chronic obstructive pulmonary disease, and Grade III-IV (NYHA) heart failure, and those with gastrointestinal bleeding who had stopped bleeding for less than 14 days after treatment or failed to stop bleeding after endoscopic variceal ligation.
* Subjects with stage C and D liver cancer (according to the Barcelona liver cancer staging criteria), or hepatocellular carcinoma (HCC) stage A/B requiring chemotherapy, intervention, surgery, or a combination of liver cancer Patients with hepatic venous cancer thrombus;
* transplant subjects
* Female subjects of childbearing age who test positive for serological pregnancy, or female subjects of childbearing age and male subjects who refuse to use contraception during the trial period or within 6 months after the last dose;
* Subjects who had participated in other clinical trials and used the investigational drug within 3 months prior to screening.
* The patient has the following laboratory test abnormalities: (1) Platelets (PLT)<30x10 ^ 9/L; Hemoglobin (HGB)<70gL; (2) Alanine aminotransferase (ALT)>5 × ULN (upper limit of normal); Aspartate aminotransferase (AST)>5 × ULN; Serum bilirubin (TBIL)>3 x upper limit of normal (ULN) ; (3) Prothrombin activity was <40%, and prothrombin time (PT) was longer than 5s; (4) Left ventricular ejection fraction (LVEF) <50%.
* Individuals who test positive for human immunodeficiency virus (HIV) antibodies; Treponema pallidum specific antibody positive and treponema pallidum non-specific antibody titer positive (unless no intervention is required during the study period assessed by the investigator);
* Other reasons the investigator considered not suitable to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2023-06-16 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-09-27 (Actual)

PRIMARY OUTCOMES:
Change from baseline in ALB | Day -1/7
  The change in albumin (ALB) was determined by calculating the difference between the value measured after the last dose (immediately after the end of dosing) and the value measured before the first dose (the mean).

SECONDARY OUTCOMES:
Improvement rate of ascites depth | Day -1/7
  Improvement of ascites depth is defined as:
  * Ascites subside in patients with baseline grade 1 ascites (none Ascites);
  * Ascites degrade in patients with baseline grade 2 ascites (ascites grade 1 or no ascites) and ascites depth drop more than 1cm;
  * Ascites depth of patients with baseline ascites grade 2 decrease by ≥ 25% and the ascites depth drop more than 1cm.
Clinical comprehensive improvement rate | Day -1/7
  The comprehensive clinical improvement was mainly based on changes in body weight and abdominal circumference. The classification and definition are:
  * Significant improvement: weight loss ≥ 1 kg, abdominal circumference improvement ≥ 2 cm;
  * Improvement: weight loss ≥ 1 kg, abdominal circumference reduction less than 2 cm; or weight loss less than 1 kg, abdominal circumference reduction ≥2 cm;
  * General improvement: abdominal circumference reduction less than 2cm and weight loss less than 1 kg;
  * Unchanged: no change or abdominal circumference reduction less than 2 cm, no change in body weight or slight increase (increase less than 1 kg); or no change in weight or loss less than 1 kg, no change in abdominal circumference or slight increase (increase less than 2cm);
  * Deterioration: Weight increase ≥ 1 kg or abdominal circumference increase ≥ 2 cm;
  * Can not judge as classified above. Improvement rate is defined as the proportion of significant improvement and Improvement subject.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No